CLINICAL TRIAL: NCT00351975
Title: A Phase I Study of PXD101 in Combination With Azacitidine (5-Aza) for Advanced Hematologic Malignancies
Brief Title: Belinostat and Azacitidine in Treating Patients With Advanced Hematologic Cancers or Other Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00146; NCI-2009-00146 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCCRC-14510A; NCI-7285; CDR0000486418; 14510A (Other: University of Chicago Comprehensive Cancer Center); 7285 (Other: CTEP); U01CA069852 (NIH); U01CA132123 (NIH); P30CA014599 (NIH); U01CA062491 (NIH); NCT00336804 (obsolete NCT alias)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2013-10

CONDITIONS: Accelerated Phase of Disease; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22;q23); MLLT3-MLL; Adult Acute Promyelocytic Leukemia With t(15;17)(q22;q12); PML-RARA; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blastic Phase; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndrome; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Philadelphia Chromosome Negative, BCR-ABL1 Positive Chronic Myelogenous Leukemia; Previously Treated Myelodysplastic Syndrome; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Disease; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Recurrence | interventions — belinostat; Azacitidine

ARMS (2):
- Arm I (chemotherapy) (Experimental): Patients receive azacitidine SC on days 1-5.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis
- Arm II (chemotherapy, enzyme inhibitor therapy) (Experimental): Patients receive azacitidine as in arm I and belinostat at the MTD IV over 30 minutes on days 1-5.
  Interventions: Drug: Belinostat; Drug: Azacitidine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Belinostat — Given IV
  Other Names: Beleodaq; PXD 101; PXD101
  Arms: Arm II (chemotherapy, enzyme inhibitor therapy)
Drug: Azacitidine — Given SC
  Other Names: 5-AC; 5-AZC; U-18496
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of belinostat when given together with azacitidine in treating patients with advanced hematologic cancers or other diseases. Belinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving belinostat together with azacitidine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of PXD101 (belinostat) when given in combination with azacitidine (when azacitidine is utilized at a dose range where its effects on cellular differentiation are known to be predominant) in patients with advanced hematologic cancers or other diseases.

SECONDARY OBJECTIVES:

I. Identify any additive or synergistic effects of this regimen on pharmacodynamic parameters, including apoptosis and re-expression of specific target genes.

II. Assess any evidence of clinical activity (complete remission, partial remission, hematologic improvement, stable disease) of this regimen in these patients.

OUTLINE: This is a dose-escalation study of belinostat followed by a randomized study.

Patients receive azacitidine subcutaneously (SC) and belinostat intravenously (IV) over 30 minutes on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of belinostat until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. After the MTD is determined, additional patients with myelodysplastic syndromes (MDS) or acute myeloid leukemia (with trilineage dysplasia or arising from MDS) are randomized to 1 of 2 treatment arms.

Arm I: Patients receive azacitidine SC on days 1-5.

Arm II: Patients receive azacitidine as in arm I and belinostat at the MTD IV over 30 minutes on days 1-5.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After receiving one course, patients randomized to arm I may crossover to receive treatment on arm II.

For patients enrolled in the randomized portion of the study, bone marrow aspirates are obtained at baseline, and after course 1 for correlative studies. Samples are examined by gene expression analysis of p15 and p21, DNA methylation of p15INK4B, and apoptosis by RT-PCR and flow cytometry. Pharmacodynamic assays are also performed.

After completion of study treatment, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of 1 of the following:

  * Relapsed or refractory acute myeloid leukemia (AML)
  * Relapsed or refractory acute promyelocytic leukemia (must have failed both tretinoin and arsenic trioxide)
  * Relapsed or refractory acute lymphoblastic leukemia
  * Secondary AML, including AML arising from antecedent hematologic diseases, such as myelodysplastic syndromes (MDS) or myeloproliferative disorders, OR therapy-related AML
  * Chronic myelogenous leukemia in accelerated or blast phase
  * Advanced phases of Philadelphia chromosome-negative (Ph-) chronic myeloproliferative disorders, as defined by ≥ 1 of the following:

    * Presence of anemia (hemoglobin < 10 g/dL and/or red blood cell transfusion dependent)
    * Presence of palpable splenomegaly
  * MDS, including chronic myelomonocytic leukemia

    * Must have intermediate or high-risk International Prognostic Scoring System (IPSS) scores (≥ 0.5)
    * Low-risk IPSS scores allowed provided ≥ 1 of the following criteria are met:

      * Hemoglobin < 10 g/dL and/or red blood cell transfusion dependent
      * Platelet count < 50,000/mm³
      * Absolute neutrophil count < 1,000/mm³
* Refractory disease OR no standard therapy exists
* Evidence of AML associated with dysplasia on bone marrow histology for elderly patients (i.e., > 60 years old) who are previously untreated and not candidates for or unwilling to undergoing induction therapy
* No known active CNS involvement with disease
* CALGB performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Bilirubin ≤ 2.0 mg/dL (unless due to Gilbert's syndrome)
* ALT ≤ 3 times upper limit of normal (unless due to disease)
* Creatinine ≤ 2 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to PXD101 or Azacitidine
* No history of allergic reactions to mannitol
* No history of dose-limiting toxicity during prior treatment with Azacitidine
* No concurrent uncontrolled illness including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude compliance with study requirements
* No marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 500 msec)
* No long QT syndrome
* No uncontrolled cardiovascular disease, including the following:

  * Severe uncontrolled hypertension
  * Uncontrolled congestive heart failure related to primary cardiac disease
  * Uncontrolled cardiac arrhythmia
  * Uncontrolled ischemic or severe valvular heart disease
  * Myocardial infarction within the past 6 months
* See Disease Characteristics
* Recovered from prior therapy
* At least 2 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas)
* At least 2 weeks since prior radiotherapy
* At least 4 weeks since prior investigational agents
* At least 24 hours since prior hydroxyurea
* At least 2 weeks since prior valproic acid
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent medication that may cause torsade de pointes
* No other concurrent anticancer therapy, including chemotherapy, radiotherapy, or biological agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of belinostat in combination with azacitidine | Course 1 (28 days)
  Graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 or 4.0.

SECONDARY OUTCOMES:
Changes in pharmacodynamic variables (target gene expression, apoptosis) | Course 1 (baseline to day 5)
  Compared between the two groups using two-sample t tests.
Association of methylation status, categorized as positive or negative, with changes in target gene expression | Baseline, days 4 or 5, and days 25-28
  Distinguished by sequence-specific polymerase chain reaction (PCR) primers. Compared using a two-sample t or Wilcoxon nonparametric test.
Clinical activity (complete remission, partial remission, stable disease, hematologic improvement) | After 4, 8, and 16 weeks
  Recorded and tabulated for both the MTD and randomized cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi Odenike, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (4):
- United States (2):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada
- Princess Margaret Hospital, Cashmere, Canterbury, New Zealand